CLINICAL TRIAL: NCT06733181
Title: The REMINDER, a Multidomain Dementia Risk Reduction Program for Older Adults Supported by Residential Care Facilities: a Feasibility Study
Brief Title: The REMINDER Program for Older Adults Supported by Residential and Daycare Facilities
Acronym: REMINDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Catarina Baptista, PhD Student, University of Coimbra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FSREMINDERRDFIORG0011881; University of Coimbra (Other: University of Coimbra)
Record Dates: First submitted 2024-11-29; First posted 2024-12-13 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Aging, Healthy; Risk Reduction; Old Age; Dementia
Keywords: Dementia risk reduction; Older adults; Multidomain programs; Residential and Daycare Facilities; Social Isolation; Loneliness
MeSH Terms: conditions — Risk Reduction Behavior; Alzheimer Disease; Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- REMINDER intervention (Experimental): The REMINDER intervention includes 20 face-to-face group sessions, each approximately 60 to 75 minutes, held twice a week over ten weeks. This program aims to optimize memory, attention, executive function, and emotional regulation while promoting lifestyle habits that protect the aging brain. The sessions include brain health education, cognitive exercises, compensatory memory strategies, training for managing personally relevant goals (with goal setting), and stress management techniques (compassion-based therapies, relaxation methods, and mindfulness). As for the structure of the sessions, each starts with a mindfulness exercise and concludes with a review of the homework assignments. Every session includes a psychoeducation component focused on a specific topic, a time for sharing and reflection, and a practical activity.
  Interventions: Other: REMINDER intervention

INTERVENTIONS:
Other: REMINDER intervention — The REMINDER intervention includes 20 face-to-face group sessions, each approximately 60 to 75 minutes, held twice a week over ten weeks. This program aims to optimize memory, attention, executive function, and emotional regulation while promoting lifestyle habits that protect the aging brain. The sessions include brain health education, cognitive exercises, compensatory memory strategies, training for managing personally relevant goals (with goal setting), and stress management techniques (compassion-based therapies, relaxation methods, and mindfulness). As for the structure of the sessions, each starts with a mindfulness exercise and concludes with a review of the homework assignments. Every session includes a psychoeducation component focused on a specific topic, a time for sharing and reflection, and a practical activity.
  Other Names: REMINDER and my brain

SUMMARY:
Dementia and mild cognitive impairment (MCI) deeply impact individuals' well-being and are expected to increase due to population aging, with global cases projected to rise to 152.8 million by 2050. Social isolation, accounting for 4% of dementia cases, emerges as a critical modifiable risk factor, particularly in institutionalized older adults, where it significantly raises dementia risk.

To address these challenges, the REMINDER program was developed as a tailored, multidomain intervention to reduce dementia risk, emphasizing social and cognitive engagement and advancing its adaptation and evaluation in Residential and Daycare Facilities (RDF). To assess the feasibility of REMINDER in older adults supported by RDF (recruitment, adherence, retention, acceptability, accessibility, and usability) and explore potential changes in cognitive and psychosocial outcomes.

DETAILED DESCRIPTION:
Implementing DRR programs in RDFs presents several unique challenges, including participant diversity in educational levels, physical and cognitive health, motivation, and logistical constraints within institutional settings. A feasibility study is essential to identify and determine how to overcome these barriers. Specifically, this study explores acceptability, accessibility, adherence, and usability to optimize the REMINDER intervention for RDF settings. By addressing these practical concerns, the feasibility trial will ensure the intervention is effective and implementable, laying the groundwork for a successful full-scale RCT that meets the needs of older adults in RDFs (resulting in an adapted version, the REMINDER4Care). By creating an engaging and well-accepted tool, we look forward to amplifying the RDF tools available to reduce the risk of dementia in their residents.

Objectives

The primary objectives of this study were as follows:

1. To evaluate the acceptance rate of RDF and participants to join the research;
2. To determine the suitability of participant eligibility criteria by estimating feasible eligibility and recruitment rates;
3. To measure participant adherence and retention through attendance rates across all intervention sessions and trends over time;
4. To assess the feasibility of the REMINDER program in clinical settings, including its acceptability, accessibility, and usability.

Secondary objectives included exploring preliminary changes in cognitive and psychosocial outcomes from baseline to post-intervention while acknowledging that the study was not powered to detect statistically significant effects.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years and older
* RDF users
* Those with elementary reading and writing skills.

Exclusion Criteria:

* Have a clinical diagnosis of dementia and/or MMSE scores below the cutoff for the presence of dementia (MMSE < 22-27, depending on education level)
* Have a psychiatric or neurological condition that impairs cognition in the long term
* Have sensory and functional deficits that compromised their participation in the neuropsychological assessment and throughout the intervention sessions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Feasibility outcomes (quantitative) | During the intervention (at the end of the sessions) and 1-week after the intervention
  Recruitment rate
Feasibility outcomes (quantitative) | During the intervention (at the end of the sessions) and 1-week after the intervention
  Adherence
Feasibility outcomes (quantitative) | During the intervention (at the end of the sessions) and 1-week after the intervention
  Retention
Feasibility outcomes (qualitative) | During the intervention (at the end of the sessions) and 1-week after the intervention
  Acceptability (with Usefulness, Satisfaction, and Ease of use (USE) questionnaire) ranges from 7 to 49, with higher scores indicating greater acceptability.
Feasibility outcomes (qualitative) | During the intervention (at the end of the sessions) and 1-week after the intervention
  Accessibility (with Usefulness, Satisfaction, and Ease of use (USE) questionnaire) ranges from 15 to 105, with higher scores indicating greater accessibility.
Feasibility outcomes (qualitative) | During the intervention (at the end of the sessions) and 1-week after the intervention
  The intervention's usability (with Usefulness, Satisfaction, and Ease of use (USE) questionnaire) ranges from 8 to 56, with higher scores indicating greater usability.

SECONDARY OUTCOMES:
Preliminary efficacy data (screening) | Screening
  Participants' sociodemographic (age in years).
Preliminary efficacy data (screening) | Screening
  Participants' sociodemographic (marital status).
Preliminary efficacy data (screening) | Screening
  Participants' sociodemographic (education level).
Preliminary efficacy data (screening) | Screening
  Participants' clinical information (presence of medical diagnosis).
Preliminary efficacy data (screening) | Screening
  Participants' clinical information (current medication).
Preliminary efficacy data (screening) | Screening
  Participants' clinical information (sensory issues).
Preliminary efficacy data (screening) | Screening
  Participants' clinical information (mobility deficits).
Preliminary efficacy data (screening) | Screening
  Participants' clinical information (substance use).
Preliminary efficacy data (screening) | Screening
  Participants' clinical information (hospitalization).
Preliminary efficacy data (screening) | Screening
  Dementia risk was assessed using the Lifestyle for BRAin health (LIBRA) score, which ranges from -2.1 to 10.6, with higher scores indicating a greater risk of developing dementia.
Preliminary efficacy data (screening) | Screening and 1-week post-intervention
  Perceived Social Isolation: This was evaluated using the Questionnaire of Perceived Social Isolation (QPSI), which is scored on a scale of 1 to 5 per item, with higher scores indicating greater perceived social isolation.
Preliminary efficacy data (screening) | Screening and 1-week post-intervention
  Global cognition was assessed using Addenbrooke's Cognitive Examination - Revised (ACE-R), a scale with scores ranging from 0 to 100, where higher scores indicate better cognitive functioning.
Preliminary efficacy data (Cognitive functions) | Baseline and 1-week post-intervention
  Episodic Memory: Measured with Word Lists I and II from the Wechsler Memory Scale-III (WMS-III), scored based on correct recalls, with higher scores reflecting better memory performance.
Preliminary efficacy data (Cognitive functions) | Baseline and 1-week post-intervention
  Processing Speed: Evaluated with the Symbol Search subtest of the Wechsler Adult Intelligence Scale-III (WAIS-III), scored by correct responses within a time limit, with higher scores representing faster processing speed.
Preliminary efficacy data (Cognitive functions) | Baseline and 1-week post-intervention
  Working Memory: Assessed with the Month Ordering task, scored by the number of correct sequences, where higher scores indicate better working memory.
Preliminary efficacy data (Cognitive functions) | Baseline and 1-week post-intervention
  Verbal Initiative: Measured with the Verbal Fluency Test (letters M, R, and alternate category), scored by the number of correct words produced, with higher scores indicating greater verbal initiative.
Preliminary efficacy data (Psychosocial/ Mental Health indicators) | Baseline and 1-week post-intervention
  Depressive Symptoms: Assessed using the Geriatric Depression Scale (GDS-30), a 30-item scale with scores ranging from 0 to 30, where higher scores indicate greater depressive symptoms.
Preliminary efficacy data (Psychosocial/ Mental Health indicators) | Baseline and 1-week post-intervention
  Loneliness: Measured with the UCLA Loneliness Scale (UCLA LS-3), the score was 20 to 80, with higher scores reflecting greater perceived loneliness.
Preliminary efficacy data (Psychosocial/ Mental Health indicators) | Baseline and 1-week post-intervention
  Social Networks: Evaluated using Lubben's Brief Social Network Scale (LSNS-6), scored from 0 to 30, where higher scores indicate a stronger social network.
Preliminary efficacy data (Psychosocial/ Mental Health indicators) | Baseline and 1-week post-intervention
  Quality of Life: This is assessed using the World Health Organization Quality of Life (WHOQOL-BREF-7), scored on a scale of 1 to 5 for each item, with higher scores indicating better quality of life.
Preliminary efficacy data (Psychosocial/ Mental Health indicators) | Baseline and 1-week post-intervention
  Life Satisfaction: This is measured using the Satisfaction with Life Scale (SWLS), scored from 5 to 25. Higher scores reflect greater life satisfaction.
Preliminary efficacy data (Perceived and performance-based functional status) | Baseline and 1-week post-intervention
  Functional capacity: This is assessed using the UPSA-2-PT (UCSD Performance-Based Skills Assessment - 2nd version), scored from 0 to 100 points, with higher scores indicating better functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology and Education Sciences, Coimbra, Portugal, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol